CLINICAL TRIAL: NCT03548818
Title: Role of Interferon-gamma 1-b (IFN-γ) on Cells of the Innate Immune System: Functional, Biochemical and Gene Expression Studies in Patients With Chronic Granulomatous Disease
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 17-1676
Record Dates: First submitted 2018-03-20; First posted 2018-06-07 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Chronic Granulomatous Disease
MeSH Terms: conditions — Granulomatous Disease, Chronic | interventions — interferon gamma-1b

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Interferon Gamma-1B — Study function and biochemistry of neutrophils off the drug for one week and then 12 hours after first dose and fourth dose.
  Other Names: None Noted

SUMMARY:
The overall goal of the study is to investigate the functional, biochemical, and gene expression effects of Interferon-gamma 1-b (IFN-γ) on the neutrophils of patients with Chronic Granulomatous Disease (CGD). The investigators hypothesize that the clinical effects demonstrated in patients with CGD treated with IFN-γ (decreased number and severity of infections) are the result of biochemical processes and upregulation of specific genes, which lead to enhanced functionality of this immune cell population.

ELIGIBILITY:
Inclusion Criteria:

* Current treatment with IFN-γ or intent to treat with this drug
* Acute infections resolved
* Subject is off treatment medications
* Women of childbearing potential must have:

  * a negative urine beta-HCG, and
  * be willing to practice two forms of effective contraception for the duration of study participation

Exclusion Criteria:

* Pregnancy,
* Breast-feeding, or
* Unwillingness to use effective contraception
* Recent vaccination (within the last fourteen days)
* Current infection or acute health condition requiring treatment
* Chronic inflammatory complications of CGD including:

  * gastric outlet or urinary tract obstruction,
  * pleuritis,
  * pericarditis,
  * inflammatory bowel disease, or
  * colitis requiring treatment.
* Un-associated chronic lung, liver, kidney, or cardiac disorders requiring active treatment

Ages: 5 Years to 60 Years | Sex: All
Age Groups: Child, Adult
Study Population: The Investigators plan to enroll children and adults, aged 5-60 years with CGD defined by functional and biochemical or genetic testing. Enrollment will be stratified by the four main variants: X-linked, gp91phox deficient patients, and autosomal recessive CGD (p47phox deficient, p67phox deficient, and p22phox deficient patients).
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2018-05-16 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Changes in Neutrophil bacterialcidal activity in patients with Chronic Granulomatous Disease (CGD) on standard treatment schedule and dose of IFN-γ in comparison to results for the patients off IFN-γ. | 1 week off drug, 12 hours after a week of treatment
  Determine changes in neutrophil function in neutrophils from patients with CGD
Changes in Gene expression as measured with RNA and affimetrics gene chips in patients with Chronic Granulomatous Disease (CGD) on standard treatment schedule and dose of IFN-γ in comparison to results for the patients off IFN-γ. | 1 week off drug, 12 hours after a week of treatment
  Determine changes in gene expression in neutrophils from patients with CGD.

SECONDARY OUTCOMES:
Differences in Neutrophil biochemical studies in patients with Chronic Granulomatous Disease (CGD) on standard treatment schedule and dose of IFN-γ in comparison to results for the patients off IFN-γ. | 1 week off drug, 12 hours after first dose of IFN-gamma; 12 hours after a week of treatment
  Determine changes in biochemical tests in neutrophils from CGD patients.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel R. Ambruso, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ambruso DR, Briones NJ, Tran AD, Sanford B, Childs C, Katz BZ, Ellison M, Johnston RB, Jones KL. Interferon-gamma 1b-induced gene expression alters neutrophil function in patients with chronic granulomatous disease. PLoS One. 2025 Sep 8;20(9):e0331657. doi: 10.1371/journal.pone.0331657. eCollection 2025. PMID 40920799